CLINICAL TRIAL: NCT02485093
Title: Comparison of Ventricular Septal Pacing With Optimized Atrioventricular (AV) Delay to no Pacing in Sinus Node Disease (SND) Patients.
Brief Title: To Pace or Not to Pace in Sinus Node Disease
Acronym: OPTIMIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008-A01266-49
Record Dates: First submitted 2013-07-26; First posted 2015-06-30 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Sinus Node Disease
MeSH Terms: conditions — Sick Sinus Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- No pacing (Active Comparator): Ventricular intrinsic conduction enhanced
  Interventions: Device: VIP
- Pacing (Experimental): Septal ventricular pacing with optimized AV delay
  Interventions: Device: Septal ventricular pacing

INTERVENTIONS:
Device: Septal ventricular pacing — Ventricular pacing must be at least 90%, from the septum and with optimized AV delay
  Arms: Pacing
Device: VIP — Ventricular pacing must be less than 10%.
  Arms: No pacing

SUMMARY:
Optimal pacing strategy for patients with SND is still unknown, although several publications in the past years demonstrated a deleterious effect of ventricular pacing. However, pacing has always been apical in these trials, and to which extent this absence of pacing is beneficial for patients with very long PR intervals is still to be found.

The aim of this study is to compare ventricular septal pacing to no pacing in patients with SND.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sinus node disease

Exclusion Criteria:

* Complete or high degree AV block
* Permanent atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2009-06; Primary Completion 2013-07 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Left Ventricular Endsystolic Diameter (LVED) | 18 months

SECONDARY OUTCOMES:
AF incidence | 18 months
Hospitalizations | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Pontchaillou - CCP, Rennes, France